CLINICAL TRIAL: NCT06941389
Title: Comparing the Effectiveness of Matched Related Donor Hematopoietic Stem Cell Transplantation to Disease Modifying Therapy in Pediatric Patients With Sickle Cell Disease.
Acronym: WeDecide
Status: Recruiting | Type: Observational
Sponsor: University of Rochester (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, John Horan, Professor - Department of Pediatrics, Hematology and Oncology (SMD), University of Rochester
Other Study IDs: BPS-2023C1-31041; BPS-2023C1-31041 (Other Grant/Funding Number: PCORI)
Record Dates: First submitted 2025-04-15; First posted 2025-04-23 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Sickle Cell Disease (SCD)
Keywords: SCD; MRD HCT; NT DMT
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- NT-DMT Cohort: This group includes 320 participants from U.S. and Canadian sites receiving non-transplant disease-modifying therapies, monitored annually over three years to assess health-related quality of life, cognitive function, disease progression, and healthcare utilization.
- MRD HCT Cohort: This group includes 160 participants from U.S. and Canadian sites receiving non-transplant disease-modifying therapies, monitored annually over three years to assess health-related quality of life, cognitive function, disease progression, and healthcare utilization.

SUMMARY:
The WeDecide study is a large observational study comparing the long-term effects of matched related donor hematopoietic stem cell transplantation (MRD HCT) and non-transplant disease-modifying therapies (NT-DMT) for pediatric patients with sickle cell disease (SCD). The study aims to assess health-related quality of life (HRQoL), cognitive function, risks, and benefits of both treatments, including survival rates, chronic complications, and organ damage prevention. With 160 children in the MRD HCT group and 320 in the NT-DMT group, aged 3-20.9 years, the study will follow participants for three years, examining factors like disease severity, treatment history, and social determinants of health. By providing a comprehensive comparison, the study seeks to inform clinical decisions and improve understanding of SCD treatment outcomes, ultimately supporting families and healthcare providers in choosing the best treatment options.

DETAILED DESCRIPTION:
The WeDecide study is a large observational study comparing the long-term effects of two treatment options for pediatric patients with sickle cell disease (SCD): matched related donor hematopoietic stem cell transplantation (MRD HCT) and non-transplant disease-modifying therapies (NT-DMT). The main goal is to understand how these treatments affect health-related quality of life (HRQoL) and cognitive function, using standard tools to measure both physical and mental health. The study also looks at risks and benefits of MRD HCT, such as the potential for chronic complications, improved survival, and prevention of organ damage.

The study includes two groups: 160 children receiving MRD HCT and 320 children receiving NT-DMT. Participants, aged 3-20.9 years, are being followed for three years. The MRD HCT group will be assessed before the transplant and then at several points post-transplant. The NT-DMT group will be assessed at the start of the study and then annually for three years.

The research also considers factors like disease severity, treatment history, and social determinants of health (such as family finances and caregiver health literacy) to better understand how these elements might influence treatment outcomes. The study tracks the use of disease-modifying therapies, as well as hospital visits and other care events, throughout the three years. It will also monitor survival rates and other important health outcomes.

This study is significant because it is the first large-scale research comparing these two treatment options for SCD in children. The results will provide essential insights into how these treatments impact long-term health and help guide clinical decisions and treatment recommendations. The goal is to help families and healthcare providers make informed decisions about the best treatment options for SCD.

The study uses advanced methods to ensure fair comparisons between the two groups by accounting for differences in their characteristics. It will also adjust for any factors that could influence the results, helping to identify meaningful differences in health outcomes between the two treatments. Ultimately, the WeDecide study aims to improve our understanding of sickle cell disease treatment and provide a foundation for future research into new therapies.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients aged between 3 and 20.9 years.
* Children diagnosed with sickle cell Anemia (HB SS or HBSB0 Thalassemia)
* For the MRD HCT group, children who are candidates for matched related donor hematopoietic stem cell transplantation (MRD HCT).
* For the NT-DMT group, children who are receiving non-transplant disease-modifying therapies (NT-DMT) for SCD.
* Participants (or their guardians) must provide informed consent to be part of the study.
* Participants must be willing to undergo the necessary assessments and follow-up visits over the 3-year study period.

Exclusion Criteria:

* Children younger than 3 years or older than 20.9 years.
* Children who do not have sickle cell anemia or related conditions.
* For the MRD HCT group, children who are not eligible for the transplant or do not have a matched related donor.
* Children who are currently enrolled in other clinical trials that might interfere with the WeDecide study.
* Children who are unable to adhere to the study protocol or follow-up requirements.

Ages: 3 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The WeDecide study includes 480 pediatric patients with sickle cell disease (SCD) from two sub-studies: Project Sickle Cure (PSC), focusing on patients receiving transplant through the Sickle Cell Transplant Advocacy Research Alliance (STAR), and the Globin Research Network for Data and Discovery (GRNDaD), a registry of patients on non-transplant disease-modifying therapies (NT-DMT) run by the National Association of Sickle Cell Centers (NASCC).
  MRD HCT Group: 160 children receiving matched related donor hematopoietic stem cell transplantation (MRD HCT) will be assessed before and at multiple post-transplant time points to evaluate long-term effects.
  NT-DMT Group: 320 children receiving non-transplant disease-modifying therapies (NT-DMT) will be assessed at study start and annually for three years to track treatment effects.
Sampling Method: Non-Probability Sample
Enrollment: 480 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2030-10-01 (Estimated); Study Completion 2030-10-01 (Estimated)

PRIMARY OUTCOMES:
Health-Related Quality of Life as Measured by the Pediatric Quality of Life Inventory (PedsQL) Generic Core Scale (Parent-Proxy Report) | Baseline, 1-year, 2-year, 3-year follow-up
  Measures physical, emotional, social, and school functioning as reported by parents.
Cognitive Function as Measured by the NIH Toolbox Cognitive Battery | Baseline, 1-year, 2-year, 3-year follow-up
  Assesses the following cognitive domains: attention, executive function, memory, language, processing speed, and working memory.

SECONDARY OUTCOMES:
Health-Related Quality of Life as Measured by the Pediatric Quality of Life Inventory (PedsQL) Generic Core Scale (Patient Reported) | Baseline, 1-year, 2-year, 3-year follow-up
  Description: Assesses self-reported physical, emotional, social, and school functioning (for age-eligible participants).
Health Related Quality of Life Using the PedsQL Sickle Cell Disease Module (Patient and Parent-Proxy Reported) | Baseline, 1-year, 2-year, 3-year follow-up
  Description: The Peds QL Sickle Cell Module assesses pain and hurt, pain impact, pain management and control, worry, emotions, treatment and communication.
Peds QL Family Impact Module (Parent Reported) | Baseline, 1-, 2- and 3-year follow-up
  Assess the burden a parent experiences. It assesses: Physical, Emotional, Social and Cognitive functioning; communication, worry, family daily activities, and family relationships.
Health Quality of Life as Measured by the Patient Reported Outcomes Measurement Information System (PROMIS, Patient and Parent-Proxy Reports) | Baseline, 1-year, 2-year, 3-year follow-up
  Assesses physical, mental and social health
The Patient Reported Outcomes Measure System (PROMIS) Pain Behavior subscale (Patient and Parent-Proxy Reports) | Baseline, 1-year, 2-year and 3-year follow-up
Number of Acute Care Visits (ED, Hospitalizations, Infusion/Clinic) | Time Points: Year 1, Year 2, Year 3
  Unit of Measure: Number of Visits per Year Description: Annual count of emergency, inpatient, or infusion center visits for acute care.
Incidence and Severity of Chronic Graft-Versus-Host Disease | Day 100, 6 months, Year 1, Year 2, Year 3
  Unit of Measure: Number of Participants with GVHD by Severity Description: Reports the GVHD occurrence in transplant recipients with severity grading.

CONTACTS AND LOCATIONS:
Locations (37):
- United States (31):
  - Children's of Alabama (MRD-HCT), Birmingham, Alabama
  - Children's of Alabama (NT-DMT), Birmingham, Alabama
  - Nemours Children's Hospital, Delaware (MRD-HCT), Wilmington, Delaware
  - Children's National Hospital (MRD-HCT), Washington D.C., District of Columbia
  - Children's Healthcare of Atlanta (MRD-HCT), Atlanta, Georgia
  - Comer Children's Hospital (MRD-HCT), Chicago, Illinois
  - Riley Children's Hospital (MRD-HCT), Indianapolis, Indiana
  - Riley's Children Hospital (NT-DMT), Indianapolis, Indiana
  - Boston Children's Hospital (MRD-HCT), Boston, Massachusetts
  - Boston Children's Hospital (NT-DMT), Boston, Massachusetts
  - Wahington Univ in St Louis (NT-DMT), St Louis, Missouri
  - Washington University in St Louis (MRD-HCT), St Louis, Missouri
  - Hackensack University Hospital (MRD-HCT), Hackensack, New Jersey
  - Roswell Park (MRD-HCT), Buffalo, New York
  - Columbia Presbytarian (NT-DMT), New York, New York
  - Cohen's Children Hospital (NT-DMT), Queens, New York
  - University of Rochester (MRD-HCT), Rochester, New York
  - University of Rochester (NT-DMT), Rochester, New York
  - Children's Hospital at Montefiore (MRD HCT), The Bronx, New York
  - Children's Hospital at Montefiore (NT-DMT), The Bronx, New York
  - UNC Children's Hospital (MRD HCT), Chapel Hill, North Carolina
  - UNC Children's Hospital (NT-DMT), Chapel Hill, North Carolina
  - Atrium Health (MRD-HCT), Charlotte, North Carolina
  - Nationwide Children's Hospital (NT-DMT), Columbus, Ohio
  - Oklahoma Children's Hospital (MRD-HCT), Oklahoma City, Oklahoma
  - Children's Hospital of Philadelphia (MRD-HCT), Philadelphia, Pennsylvania
  - St Jude Children Hospital (NT-DMT), Memphis, Tennessee
  - St. Jude Children's Research Hospital (MRD-HCT), Memphis, Tennessee
  - Texas Children's Hopsital (NT-DMT), Houston, Texas
  - Texas Children's Hospital (MRD-HCT), Houston, Texas
  - UT San Antonio (NT-DMT), San Antonio, Texas
- Canada (6):
  - Alberta Children's Hospital (NT-DMT), Calgary, Alberta
  - Alberta Children's Hospital (MRD-HCT), Calgary, Alberta
  - British Columbia Children's Hosptial (MRD HCT), Vancouver, British Columbia
  - HSC Winnipeg Children's Hospital/University of Manitoba (MRD-HCT), Winnipeg, Manitoba
  - The Hospital for Sick Children (MRD-HCT), Toronto, Ontario
  - Universite de Montreal / Ste Justine (MRD HCT), Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No